CLINICAL TRIAL: NCT04035291
Title: Effectiveness of Family Collaborative Physiotherapy Programs With High-risk Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hatice Adıgüzel, Principal Investigator, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sanko U
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy; Infant, Newborn, Disease; Infant, Small for Gestational Age; Infant Asphyxia; Infant, Very Low Birth Weight; Infant of Diabetic Mother; Infant, Premature, Diseases; Infant Development
Keywords: Family Collaboration,; high risk of CP; physiotherapy
MeSH Terms: conditions — Cerebral Palsy; Disease; Infant, Premature, Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Infants will be divided into two groups according to prenatal risk factors (maternal age, intrauterine growth retardation, chronic diseases etc.) by random minimization method and taken into 2 different physiotherapy programs. As the control group, the group participating in the evaluations stating that they cannot participate in the treatment without any intervention will be taken.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All of the interventions will be shown to the infants' (participants') parents by the investigator physiotherapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interventional (Active Comparator): The first group (n = 25) will be asked to apply the physiotherapy program by the family at home that includes the principles of therapeutic handling-holding-positioning of NDT principles, starting at the third month for 8 weeks. And It will last for at least 45 minutes, 3 days a week. Family education will be evaluated after 4 weeks and improvements will be made in accordance with the motor development of the infant. The program will be implemented by families for 8 weeks.
  Interventions: Other: exercise
- Experimental (Experimental): In the second study group (n = 25), family collaborative physiotherapy program will be applied by the family. This program will start from the postterm third month, and will include family trainings based on the goal-oriented active motor learning model of the baby in an 8-week in enriched environment and to include holding-carrying-positioning trainings in daily routines. Also it will last for at least 45 minutes, 7 days a week. All members of the family will be included in the family trainings and home visits will be made at 2-week intervals. Families will be encouraged to apply the physiotherapy processes of their babies in their natural environment at every moment of their daily routines (feeding, carrying on lap, gas extraction, changing the bed, sleeping, waking time, shopping moment, playing games etc.).
  Interventions: Other: exercise
- control (No Intervention): In the third study group, families who are out of town or who cannot participate in the treatment program for other reasons will be included in the evaluations.

INTERVENTIONS:
Other: exercise — exercises,play therapy models and positioning, handling and holding principles for babies, daily routins
  Arms: Experimental; Interventional

SUMMARY:
High risk infant is defined as infant with a negative history of environmental and biological factors, which can lead to neuromotor development problems. It is a heterogeneous group of premature infants born under thirty-seven weeks of age, with infants with low birth weight, term or developmental retardation for various reasons. Therefore, preterm infants with low birth weight can survive with a neurological sequelae such as cerebral palsy (CP), epilepsy, hearing and vision loss, mental retardation, speech and speech problems, and learning difficulties. The clinical diagnosis of CP, which can be observed in high-risk infants, is based on the combination of some neurological and clinical signs. High-risk of infant follow-up programs provide guidance for the treatment of neurodevelopmental delays and deterioration in terms of early development. Three methods with the best predictable validity that can determine CP before the adjusted age of 5-month is Magnetic Resonance Imaging (MRI), Prechtl's Assessment of General Movements (GMs), Hammersmith Infant Neurological Evaluation. In recent years, the diagnosis of high-risk of CP can be detected at 3 months with predictive validity and reliability by evaluating the quality of GMs. GMs are now considered the gold standard for early detection of CP because of its high sensitivity and specificity than MRI, cranial US and neurological evaluations. It was also found that cognitive or language skills may be inadequate in school age in patients with inadequate movement character and in the same postural patterns according to age, although GMs are normal. So new clinical care guidelines and new intervention research for infants with CP under the age of 2, needed to have been shown. High-risk infants who are thought to have developmental disorders need early intervention, but it is not yet known which interventions are more effective. In the literature, although interventions are generally shown to have a greater impact on cognitive development, their contribution to motor development cannot be fully demonstrated. The effectiveness of physiotherapy programs in the diagnosis and treatment of CP has not been clarified in the past years as a silent period. Therefore, studies involving early physiotherapy programs are needed in infants at high risk for CP.

DETAILED DESCRIPTION:
High-risk infants who are thought to have developmental disorders need early intervention, but it is not yet unknown which interventions are more effective. In the literature, although interventions are generally shown to have a greater impact on cognitive development, their contribution to motor development cannot be fully demonstrated. Early physiotherapy and rehabilitation in CP includes approaches starting from the neonatal period up to 24 months. The main aim is to gain normal functional movements and to provide normal sensory input by using the rapid learning ability resulting from brain plasticity. Thus, it is aimed to reach the most independent level in terms of physical, cognitive, psychological and social aspects within the physiological and anatomical deficiencies and environmental limitations of the child. In the literature, there are studies including interventions to preterm infants with high risk for developmental disorder. However, although the number of samples in the studies is high, there is insufficient information about the rate of CP development. The effectiveness of physiotherapy programs in the diagnosis and treatment of CP has not been clarified in the past years as a silent period. Therefore, studies involving early physiotherapy programs are needed in infants at high risk for CP. Preterm infants have been shown to have difficulty in most functional areas due to lower academic success, welfare and productivity. These difficulties may arise in childhood and adolescence due to brain damage and structural changes. The stress of being away from mother contact has been proven in human and experimental animal studies. Physical and emotional environment modifications of the babies in the incubator environment can also reduce stress. Parent-centered trainings that will increase sensitivity in the intensive care unit by reducing stresses in the brain in terms of early intervention; it has been shown to have positive reflections on motor and cognitive development in the short term. In the literature, it has been shown that the specific motor education programs and the interventions that parents learn how to support the development of their babies are the most important ways to increase the cognitive development of infants at high risk by reducing motor disorders. It is essential to force babies to produce motor behavior on their own, knowing the limits of motor behavior. It is then essential to ensure that babies continue this activity and to use stimulations for this. There may be positive developmental outcomes in physiotherapy models such as COPCA, where parental coaching is performed. However, further studies are needed in this area. These physiotherapy approaches are necessary to reduce the risk for motor and cognitive development and to achieve normal motor development. In particular, the motor and cognitive development of infants at high risk of CP should be monitored. In the literature, an early rehabilitation model that includes physiotherapy in family routines has shown that some problems with high risk of infants need to be focused on by early physiotherapy approach. In our study, the effectiveness of family education and family cooperative physiotherapy programs in accordance with NDT-based neurodevelopmental treatment principles applied to infants with high risk of CP will be examined. The effect of physiotherapy methods applied to infants on motor and cognitive development levels will be investigated according to the risk factors and physiotherapy model. In addition, the effects of physiotherapy programs on the possibility of decreasing the symptoms of CP or preventing the development of CP will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Periventricular hemorrhage, patients with intracranial hemorrhage grade 2, 3, 4, cystic periventricular leukomalacia, Stage 3 hypoxic ischemic encephalopathy, Neonatal bilirubin encephalopathy (kernicterius), perinatal stroke, perinatal asphyxia, babies with hydrocephalus
* Chronic pulmonary disease Infants with dysplasia and long-term O₂ support
* Preterm infants with sepsis, necrotizing enterocolitis (NEC), infantile apnea, cerebral malformation due to gram negative bacteria
* Patients with a low Apgar score of 5 minutes (3 and less), multiple births (twins, triplets) diagnosed with intrauterine growth retardation, preterm infants with premature retinopathy (ROP)
* Infants with prolonged severe hypoglycemia and hypocalcemia
* Surgical conditions such as diaphragmatic hernia or tracheoesophageal fistula
* Infants younger than gestational age (Small for Gestational Age, SGA, smaller than 3rd percentile) or older than gestational age (Large for Gestational Age, LGA, greater than 97th percentile)
* Babies receiving mechanical ventilation for more than 24 hours
* Babies less than 32 weeks of gestation and born under 1500 g

Exclusion Criteria:

* Infants with congenital malformation (Spina Bifida, Congenital Muscular Torticollis, Arthrogriposis Multiplex Congenita etc.)
* Infants diagnosed with metabolic and genetic diseases (Down Syndrome, Spinal Muscular Atrophy, Duchenne Muscular Dystrophy etc.)
* Infants still intubated and mechanical ventilator dependent at postterm 3 months

Ages: 24 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change of Bayley Scales of Infant and Toddler Development (Bayley-III) score | 3th and 6th months (before and after intervention)
  measures cognitive, language, motor, socio-emotional and adaptive behaviors of children between 0-42 months.High scores shows better development.
Change of Hammersmith infant neurological examination test score | 2, 3 and 6th months
  The use of the HINE optimality score and cut-off scores provides prognostic information on the severity of motor outcome. The HINE can further help to identify those infants needing specific rehabilitation programs.High scores shows better developmental stage.

SECONDARY OUTCOMES:
Change of the General Movement Assessment (GMs) | Maximum 2 times in the preterm period, 2 times until the 10th week, postterm 10th week-24. 4-6 camera recordings will be taken for 5 minutes, 2 times per week.
  Gms can identify neurological issues predictive of cerebral palsy and other developmental disabilities.GMs videos around 3 months of age (12-16 weeks corrected age) provide the most predictive information about the likelihood risk of cerebral palsy. Ther isn't maximum or cut off scores.Movements are noted as observed/or not. Also quality of fidgety movements are scored as low or high quality.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Adıgüzel, PhD cd., Principal Investigator — Sanko University
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)